CLINICAL TRIAL: NCT06616870
Title: Study of the Predictive and Prognostic Role of Pharmacogenetic and Radiogenic Variants on the Response to Neoadjuvant Chemoradiation Therapy in Patients With Locally Advanced Rectal Cancer
Acronym: IGLarc
Status: Not yet recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-77
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In locally advanced rectal cancer the pathological complete response (pCR) to neoadjuvant chemoradiation therapy (nCRT) is associated with a favourable long-term prognosis. The identification of markers predictive of response to therapy would therefore optimise treatment by allowing personalised therapy. It has been shown that the genetic profile of the patient could influence the activation of the immune system in combination with chemoradiation therapy in targeting tumour cells. In addition, genetic features of molecular pathways correlated with response to chemoradiotherapy, may in turn affect the probability of a good response to treatment in these patients, but also the occurrence of adverse events. The main objective of the study is to define the role of genetic markers related to immune system activation and other molecular pathways in predicting the complete pathological response to preoperative chemoradiation therapy in patients with locally advanced rectal cancer.

ELIGIBILITY:
Eligibility criteria:

1. histologically confirmed diagnosis of primary resectable LARC;
2. confirmed absence of distant metastases;
3. ≥18 years old;
4. stage of disease T3-T4 and N0-N2;
5. performance status (World Health Organisation) 0-2;
6. normal bone marrow, kidney and liver function;

Exclusion Criteria:

1. evidence of secondary tumour
2. inadequate liver function (bilirubin >1.5 times the normal range, ALT and AST >2 times the normal range);
3. inadequate renal function (creatinine >1.5 times the upper limit of normal range);
4. Major concomitant systemic diseases that contraindicate surgery;
5. significant cardiovascular disease (heart failure, acute myocardial infarction within the last year, active angina, cardiac arrhythmia to be treated, uncontrolled hypertension)
6. systemic disease contraindicating radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically confirmed diagnosis of primary resectable LARC
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2024-10-03 (Estimated); Primary Completion 2029-10-03 (Estimated); Study Completion 2029-10-03 (Estimated)

PRIMARY OUTCOMES:
Defining the predictive role of rare (MAF<1%) and very rare genetic variants (MAF<0.1%) in the SMAD3 and IL-17F genes, implicated in nCRT-mediated activation of the immune system on the pathological tumour response to nCRT in LARC. | up to 5 years
  Relation between rare and very rare genetic variants and pathological tumour response will be assessed with logistic regression analysis and data will be reported as odds ratio and relative confidence interval

SECONDARY OUTCOMES:
Plasma levels of IL-17F and SMAD3 proteins during treatment to be correlated with the genetic characteristics | up to 5 years
  Mean difference between subgroup of patients with different genetics characteristics
Plasma levels of IL-17F and SMAD3 proteins during treatment and tumour response | up to 5 years
  Relation between plasma levels of IL-17F and SMAD3 proteins and pathological tumour response will be assessed with logistic regression analysis and data will be reported as odds ratio and relative confidence interval
Plasma levels of IL-17F and SMAD3 proteins during treatment and prognosis of the tumour. | up to 5 years
  Relation between plasma levels of IL-17F and SMAD3 and disease-free survival (DFS) defined as time between enrollment and objective tumor progression using Kaplan Meyer method
Identify further genetic markers of pathological tumour response | up to 5 years
  Relation between selected genetic markers and pathological tumour response will be assessed with logistic regression analysis and data will be reported as odds ratio and relative confidence interval
Define the role of the same genetic polymorphisms on disease-free survival | up to 5 years
  Relation between selected genetic markers and disease-free survival (DFS) defined as time between enrollment and objective tumor progression using Kaplan Meyer method
Define the role of the same genetic polymorphisms on overall survival of patients | up to 5 years
  Relation between selected genetic markers and overall survival (OS) defined as time between enrollment and death from any cause using Kaplan Meyer method
Define the role of the same genetic polymorphisms on the risk of developing severe treatment toxicities | up to 5 years
  Relation between genetic variants and severe treatment toxicity will be assessed with logistic regression analysis and data will be reported as odds ratio and relative confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Erika Cecchin, PhD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy